CLINICAL TRIAL: NCT03495193
Title: Impact of a Novel Exercise Intervention on Executive Function and Sleep in Patients With Parkinson's Disease
Brief Title: Impact of Exercise in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Parkinson's Disease Foundation (Other)
Responsible Party: Principal Investigator, Amy Amara, MD, Associate Professor of Neurology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-170324012
Record Dates: First submitted 2018-03-27; First posted 2018-04-11 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized, controlled, interventional study to investigate the impact of a novel exercise intervention on executive dysfunction (Aim 1) and objective sleep outcomes (Aim 2) in patients with PD. Thirty participants with idiopathic PD will be recruited from the University of Alabama at Birmingham (UAB) Movement Disorders Center and randomized (1:1) to one of two groups (15 per group): exercise intervention (Ex) group or no-exercise (no-Ex) control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): Subjects randomized to the exercise training group will complete 16 weeks of exercise training. Exercise training will be performed 3x/week.
  Interventions: Other: Exercise training
- No Exercise Group (Active Comparator): Subjects randomized to the no-Ex group will receive a handout with tips for improving sleep hygiene. Additionally, study staff will provide the title page for a book on sleep relaxation techniques that is recommended for persons with sleeping difficulty.
  Interventions: Behavioral: Sleep hygiene

INTERVENTIONS:
Other: Exercise training — Exercise training will be performed 3x/week. After 2 sessions, training volume and intensity will progress over the first 4 sessions ramping up the number of sets to increase the volume. The full volume prescription will consist of: 1) 5 movements to improve strength and muscle mass (leg press, knee extension, chest press, overhead press, pull down), 3 sets each of 8-12 repetitions (~30 total repetitions); 2) trunk exercises to improve postural stability (trunk extension and flexion); 3) 3-4 bodyweight exercises (selected from a menu) to improve power and balance (e.g. step up, squat, jump squat, lunge, side lunge, push-up, assisted pull-up, assisted dip). Bodyweight movements will be modified as necessary to match abilities.
  Arms: Exercise Group
Behavioral: Sleep hygiene — Subjects randomized to the no-exercise group will receive a handout with tips for improving sleep. Additionally, study staff will provide the title page for a book on sleep relaxation techniques that is recommended for persons with sleeping difficulty. Dr. Amara will review the sleep tips with the subjects and make recommendations for improving current sleep habits. Subjects will be contacted by telephone every 4 weeks during the 16-week intervention period.
  Arms: No Exercise Group

SUMMARY:
The goal of this research is to identify an intervention that will improve cognition and sleep in persons with PD.

DETAILED DESCRIPTION:
Persons with Parkinson's disease (PD) often experience non-motor symptoms such as cognitive dysfunction and sleep problems. These symptoms can be more disabling than the motor symptoms of PD. Medications are often not effective for treating these non-motor symptoms or can have unwanted side effects. Non- medication treatments such as exercise are known to improve the motor symptoms of PD, but the effect of exercise on cognition and sleep has not been fully explored. This study investigates the impact of 16 weeks of supervised exercise, 3 times per week, compared to no-exercise over the same duration, on cognition and sleep dysfunction. Participants will be evaluated with cognitive tests and sleep studies before and after 16-weeks to determine the impact of this exercise intervention. The goal of this research is to identify an intervention that will improve cognition and sleep in persons with PD.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of idiopathic PD, based on the presence of bradykinesia as well as rest tremor and/or rigidity;
* Hoehn and Yahr stage 2-3;
* age ≥ 45;
* on stable medications for at least 4 weeks prior to study entry;
* Participants must have Montreal Cognitive Assessment (MoCA) score ≥ 18;
* No contraindications to an exercise program, based on the Physical Activity Readiness Questionnaire (PAR-Q), resting physical examination, and 12-lead electrocardiogram.

Exclusion Criteria:

* features suggestive of atypical Parkinsonism (cerebellar signs, supranuclear gaze palsy, prominent autonomic failure, or prominent upper motor neuron signs);
* secondary Parkinsonism (multiple strokes with stepwise progression of Parkinsonism, neuroleptic treatment at time of diagnosis, or multiple head injuries);
* inability to walk without a cane or walker;
* regular participation in an exercise program in the past 6 months;
* presence of deep brain stimulator; and
* untreated sleep apnea.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Executive function (Stroop inhibition, Trails B-A, Controlled oral word association) | changes from baseline to week 16
  Changes in executive function will be measured by a change in a composite executive function score calculated from the mean of z-scores for Stroop inhibition, Trails B-A, and COWA.
Sleep Efficiency | changes from baseline and week 16
  Change in sleep efficiency (the number of minutes asleep divided by the number of minutes in bed) between the baseline nocturnal polysomnography to the post-16 weeks of intervention nocturnal polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886